CLINICAL TRIAL: NCT04311450
Title: Behavioral Weight Loss Treatment for Individuals With Food Addiction
Acronym: FA Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2000027229
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Food Addiction; Overweight and Obesity; Weight Loss
MeSH Terms: conditions — Food Addiction; Overweight; Obesity; Weight Loss | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss (Experimental): Behavioral: Participants randomized assigned to this arm will received 12 weeks of Behavioral Weight Loss (BWL) counseling.
  Interventions: Behavioral: Behavioral Weight Loss (BWL) counseling
- Waitlist Control (No Intervention): Waitlist Control: Participants assigned to this arm will attend follow-up visits to control for the effect of time. Following completion of post-treatment assessment participants in the waitlist control group will be offered an abbreviated BWL treatment.

INTERVENTIONS:
Behavioral: Behavioral Weight Loss (BWL) counseling — This therapy is a weekly treatment which focuses on making gradual and modest lifestyle changes with goals of establishing regular patterns of eating, setting weekly goals, decreasing caloric intake, developing coping skills, and increasing physical activity.
  Arms: Behavioral Weight Loss

SUMMARY:
The purpose of this research study is to examine how well an existing weight loss treatment works for individuals with food addiction. Treatment will consist of a preliminary 12-week RCT pilot of the feasibility and effectiveness of behavioral weight loss (BWL) compared to a waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-50 kg/m2
* Meets criteria for Food Addiction (based on the self-report score from the Yale Food Addiction Scale)
* Available for the duration of the treatment (3 months)
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* Availability of internet to participate in study interventions (i.e., electronic SMART scales)

Exclusion Criteria:

* Co-existing psychiatric condition that requires hospitalization or more intensive treatment (e.g., bipolar mood disorders, psychotic illnesses, severe depression).
* Reports active suicidal or homicidal ideation
* Current anorexia or bulimia nervosa
* Endorsing current or history of heart trouble/chest pain.
* Breast-feeding or pregnant, or planning to become pregnant during the study.
* History of stroke or myocardial infarction.
* Current or recent (within 12 months) drug or alcohol dependence
* Currently receiving effective treatment for eating or weight loss, including individual who received bariatric surgery within the past five years
* Currently participating in another clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Weight (e.g., change in percent weight loss) | Up to 12 weeks
Food addiction (change in food addiction scores) | Up to 12 weeks
  Yale Food Addiction Scale scores will be assessed by self-report (range of scores 0-7, higher score reflect greater food addiction symptoms)

SECONDARY OUTCOMES:
Food Craving (change in food craving scores) | Up to 8 weeks
  Food Craving Inventory scores will be assessed by self-report (range of score 0-185, higher scores reflect greater food cravings).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States